Mid- and long-term surgical and oncological outcomes of total laparoscopic gastrectomy for gastric cancer: A prospective study. November 25, 2020

## STUDY PROTOCOL

- 1. Background and current status of the issue: the laparoscopic approach for gastric carcinoma (GC) is being increasingly implemented by digestive surgeons. Although recent evidence suggests that this surgical approach is associated with improvements in short-term outcomes, mid- and long-term outcomes have not been well studied.
- 2. Study justification: laparoscopic gastrectomy for GC is widely employed in eastern Countries. But there is a lack of data on its use and results in Western countries, where the incidence of this pathology is lower.

but there is much less information on its use in western countries

- 3. Goals: This study aimed to evaluate the mid- and long-term outcomes of laparoscopic gastrectomy (LG) with D1-D2 lymph node dissection for all stages of GC in a western country.
- 4. General objectives: to establish a program for the laparoscopic treatment of GC.
- 5. Specific objectives: determine the short, medium and long-term results of the program.
- 6. Hypothesis: the results should be similar to those reported by eastern centers.
- 7. Methodology: prospective observational study.
- 8. Reference and study population: patients diagnosed of GC and fits for surgery.
- 9. Inclusion criteria:
- a. Patients diagnosed with gastric adenocarcinoma and operated by a laparoscopic approach.
- b. Acceptance the proposed technical procedure by the patient.
- c. No anesthetic contraindication for the laparoscopic technique.
- 10. Exclusion criteria:
- a. Patients lost to follow-up.
- b. Patients unfit for surgery.
- c. Palliative surgery.
- d. T4b lesions or gastric neoplasms other than adenocarcinoma
- 11. Sample size: 100-150 cases.
- 12. Variables:
- a. Demographic data.
- b. Operative morbidity and mortality.
- c. Disease-free survival at 3, 5, and 10 years.
- d. Overall survival at 3, 5 and 10 years.
- e. Neoadjuvant and / or adjuvant treatment.
- 13. Data collection and information sources: The data obtained will be collected in an ANONYMOUS database and guarded by the main researcher and the researchers signing the project, respecting at all times Organic Law 15/1999, of December 13, on the Protection of Personal Data.

14. Analysis of data: The statistical program IBM SPSS Statistics 25.0 will be used. A descriptive analysis of the collected data will be carried out, based on survival or mortality during the follow-up period and, later, it will be made with a Cox regression, a univariate and multivariate analysis, with the in order to determine the risk factors for mortality at one year, three, five and ten years of follow-up